CLINICAL TRIAL: NCT07017257
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation in Patients With Persistent Post-concussion Symptoms: a Randomized Double-blind Controlled Trial
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation for Persistent Post-concussion Symptoms
Acronym: taVNS-PPCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: University Hospital Sart Tilman, Liege (Unknown)
Responsible Party: Principal Investigator, Aurore Thibaut, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-373
Record Dates: First submitted 2025-05-08; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Persistent Post-concussive Symptoms
Keywords: Vagus nerve stimulation; Transcutaneous electrical nerve stimulation; Non-invasive brain stimulation; Persistent post-concussive symptoms; High-density EEG

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active taVNS (Experimental): Patients will undergo 15 sessions of 30-min active taVNS applied to the cymba conchae of the left ear. Clinical assessments-including symptom severity questionnaires and neuropsychological tests-along with neurophysiological recordings (hd-EEG and electrocardiography) will be conducted on the first (S1) and final (S15) days of the intervention. The remaining 13 sessions (S2-14) will be self-administered by patients at home.
  To monitor safety, participants will report any side effects after each session.
  To monitor adherence, the device will record the time and duration of each stimulation session. Blinding efficacy will be evaluated at the end of the intervention by asking participants to indicate whether they believe they received active or sham stimulation, and to rate their confidence in that response.
  A follow-up assessment will occur one month after the intervention, during which symptom severity questionnaires will be administered via a phone interview.
  Interventions: Device: Active taVNS
- Sham taVNS (Sham Comparator): Patients will undergo 15 sessions of 30-min sham taVNS applied to the cymba conchae of the left ear. Clinical assessments-including symptom severity questionnaires and neuropsychological tests-along with neurophysiological recordings (hd-EEG and electrocardiography) will be conducted on the first (S1) and final (S15) days of the intervention. The remaining 13 sessions (S2-14) will be self-administered by patients at home.
  To monitor safety, participants will report any side effects after each session.
  To monitor adherence, the device will record the time and duration of each stimulation session. Blinding efficacy will be evaluated at the end of the intervention by asking participants to indicate whether they believe they received active or sham stimulation, and to rate their confidence in that response.
  A follow-up assessment will occur one month after the intervention, during which symptom severity questionnaires will be administered via a phone interview.
  Interventions: Device: Sham taVNS

INTERVENTIONS:
Device: Active taVNS — Patients will receive active taVNS for 15 consecutive days, with each session lasting 30 minutes. The stimulation will target the cymba conchae of the left ear and will consist of alternating 30-second on and 30-second off periods. The current intensity will range from 1 to 3 mA, adjusted to the patient's pain threshold, with a pulse width of 250 μsec and a frequency of 25Hz.
  Arms: Active taVNS
Device: Sham taVNS — Patients will receive sham taVNS for 15 consecutive days, with each session lasting 30 minutes. The stimulation will target the cymba conchae of the left ear and will consist of alternating 30-second on and 30-second off periods. The current intensity will be fixed at 100 µA, with a pulse width of 250 μsec and a frequency of 25 Hz.
  Arms: Sham taVNS

SUMMARY:
Persistent post-concussive symptoms (PPCS) affect a significant proportion of individuals following a concussion, leading to debilitating impacts on their quality of life and work capacity. Currently, effective treatments for PPCS are limited, despite their lasting and debilitating impact. Transcutaneous auricular vagus nerve stimulation (taVNS), a non-invasive neuromodulation technique, holds promise as a therapeutic option by leveraging the bottom-up modulation of brain activity via the auricular branch of the vagus nerve. This study aims to evaluate the neurophysiological and clinical effects of taVNS on brain activity and symptomatology in patients with PPCS through a randomized, controlled, double-blind trial.

DETAILED DESCRIPTION:
PPCS occur in 30-50% of individuals following a concussion and can persist for months, causing somatic complaints (e.g., headaches and dizziness), cognitive impairments (e.g., memory and concentration issues), emotional disturbances (e.g., anxiety and depression), and sleep disorders. Despite their long-term consequences, effective treatments for PPCS remain scarce. Transcutaneous auricular vagus nerve stimulation (taVNS) is a promising non-invasive technique that stimulates the auricular branch of the vagus nerve to induce bottom-up effects on brain activity, potentially alleviating PPCS.

This randomized, controlled, double-blind clinical trial will evaluate the cumulative and direct neurophysiological and clinical effects of taVNS (tVNS Technologies GmbH, Germany) in 48 patients aged 18 to 65 years who experienced a diagnosed concussion between 4 weeks and 1 year prior to enrollment and suffer from PPCS. Participants will be randomized to either an active taVNS group or a sham stimulation group.

Patients will undergo a total of 15 taVNS sessions over two weeks, including two visits at the University Hospital of Liège (first and last session) and 13 self-administered sessions at home. Symptom severity, including headaches, depression, anxiety, sleep disturbances, and overall quality of life, will be measured using validated questionnaires, while cognitive function (i.e., attention, working memory, executive functions) will be assessed through neuropsychological tests. Additionally, electroencephalographic (EEG) and electrocardiogram (ECG) recordings will be used to measure changes in brain activity and heart rate, respectively, focusing on alterations in power spectral density and functional connectivity patterns that may correlate with clinical improvements.

Follow-up assessments will occur one-month post-intervention via a phone call to collect questionnaires assessing symptom severity and quality of life.

This protocol aims to provide robust evidence on the efficacy and mechanisms of taVNS for PPCS while advancing our understanding of the neurophysiological changes associated with this therapeutic approach.

Interim analyses will be conducted after the inclusion of 24 patients to evaluate preliminary data. These analyses will also allow for adjustments to the sample size, if necessary, to maintain the study's statistical power.

Patients who did not complete 80% of the sessions (12 sessions) will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65;
* Between 4 weeks and 1-year post-diagnosis of a concussion;
* Score equal or above 16 on the Rivermead Post-Concussion Questionnaire;
* Intact skin at the electrode site.

Exclusion Criteria:

* History of chronic neurological or psychological disorders (still untreated 6 months preceding inclusion);
* Pregnancy or breastfeeding;
* Presence of an active implant (e.g., pacemaker, cochlear implant);
* History of myocardial infarction or cardiac arrhythmia;
* Excessive alcohol consumption (> 14 drinks per week) and/or drug (> 1x/week) use within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Effects of taVNS on symptom severity in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  The investigators will evaluate the effects of taVNS on the severity of PPCS, as measured by the Rivermead Post-Concussion Questionnaire (RPQ). The RPQ consists of 16 items scored on a 5-point Likert scale (0 = not experienced at all, 4 = severe problem). Total scores range from 0 to 64, with higher scores indicating worse symptom severity. The RPQ will be administered at four time points: baseline, mid-treatment, post-intervention, and one-month follow-up.
Effects of taVNS on brain activity in patients with PPCS | From enrollment to the end of the treatment at 2 weeks.
  The investigators will assess the effects of taVNS on brain activity using electroencephalography (EEG). Specific metrics analyzed will include:
  * Power spectral density across frequency bands: delta (0.5-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and gamma (30-45 Hz).
  * Functional connectivity patterns across cortical regions based on EEG coherence or phase-locking value.
  These parameters will be extracted from EEG data collected before and after the first and final taVNS sessions.

SECONDARY OUTCOMES:
Effects of taVNS on cognitive functions in patients with PPCS | From enrollment to the end of the treatment at 2 weeks.
  Cognitive performance will be assessed using the Test of Attentional Performance (TAP v2.3.1). Individual domain scores will be reported according to test-specific metrics. This assessment will be performed at baseline and after the intervention.
Effects of taVNS on verbal memory in patients with PPCS | From enrollement to the end of the treatment at 2 weeks.
  The Rey Auditory Verbal Learning Test (RAVLT) will be performed to evaluate verbal memory. This test will be conducted at baseline and post-intervention. Individual domain scores will be reported. This assessment will be performed at baseline and after the intervention.
Effects of taVNS on heart rate variability in patients with PPCS | From enrollment to the end of the treatment at 2 weeks.
  The investigators will assess heart rate variability (HRV) using electrocardiogram (ECG) recordings. Heart rate variability measurements will be performed before and after the first and final taVNS sessions.
Effects of taVNS on headaches in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  The Headache Impact Test (HIT-6) will be used to evaluate the severity of headaches. Scores range from 36 to 78, with higher scores indicating worse impact. This questionnaire will be administered at three time points: baseline, post-intervention and at one-month follow-up.
Effect of taVNS on sleep quality in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) (score range: 0-21; higher scores = worse sleep quality). This questionnaire will be administered at baseline, post-intervention, and follow-up.
Effects of taVNS on daytime sleepiness in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS) (score range: 0-24; higher scores = greater daytime sleepiness). This questionnaire will be administered at baseline, post-intervention, and follow-up.
Effects of taVNS on sleep changes in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  Changes in sleep will be assessed using the Sleep and Concussion Questionnaire (SCQ) (score range: 0-36; higher scores = greater severity and frequency of sleep disturbances). This questionnaire will be administered at baseline, post-intervention, and follow-up.
Effects of taVNS on depressive symptoms in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  Depressive symptoms will be evaluated using the Beck Depression Inventory (BDI-II) (score range: 0-63; higher scores = more severe depression). This questionnaire will be administered at baseline, post-intervention, and follow-up.
Effects of taVNS on anxiety symptoms in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  Anxiety symptoms will be evaluated using the Beck Anxiety Inventory (BAI) (score range: 0-63; higher scores = more severe anxiety) This questionnaire will be administered at baseline, post-intervention, and follow-up.
Effects of taVNS on quality of life in patients with PPCS | From enrollment to the end of the study at 6 weeks (including follow-up).
  The Quality of Life after Brain Injury Questionnaire (QOLIBRI) will be used to assess quality of life. The total score ranges from 0 to 100, with higher scores indicating better quality of life. This questionnaire will be administered at three time points: baseline, post-intervention and at one-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lejeune, MD, PhD, Principal Investigator — NeuroRehab & Consciousness Clinic, Neurology Department , University Hospital of Liège; Aurore Thibaut, PT, PhD, Principal Investigator — NeuroRecovery Lab, GIGA-Consciousness, GIGA Institute, University of Liège
Locations (1):
- University Hospital of Liège, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided